CLINICAL TRIAL: NCT00565305
Title: Quality of Life and Immunity During Breast Cancer Treatment
Brief Title: Healing Touch, Quality of Life, and Immunity During Breast Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Lutgendorf, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 200305053
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: Healing Touch; NK cytotoxicity; cytokines; fatigue
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healing Touch (Experimental): Healing Touch + Standard Treatment Healing Touch treatments daily following standard Radiation Therapy. Standard radiation therapy is part of their medical care and is not administered as part of this study. Protocol of 4 HT techniques will be used including Pain Drain, Chakra connection, Magnetic Unruffling, and Mind Clearing. Treatments will be approximately 20-30 minutes.
  Interventions: Behavioral: Healing Touch; Radiation: Standard Treatment
- Usual Care (Active Comparator): Standard Treatment. These patients receive usual medical care but no additional intervention. Standard treatment is not administered as part of this study but as part of their medical treatment.
  Interventions: Radiation: Standard Treatment

INTERVENTIONS:
Behavioral: Healing Touch — Healing Touch (HT) is a non-invasive therapeutic approach to healing which describes its mode of action as using touch to modulate the patient's energy system. The goal of HT is to restore harmony and balance in the patient's energy system to assist the person to self-heal.88 Healing Touch, as used here, refers to the techniques taught in Mentgen's standardized curriculum of Healing Touch offered through Healing Touch International and endorsed by the American Holistic Nurse's Association
  Arms: Healing Touch
Radiation: Standard Treatment — 4-6 cycles of cytotoxic chemotherapy followed by 5040 cGy of external beam whole breast radiotherapy in 28 fractions usually followed by a boost of 1000-1600 cGy

SUMMARY:
The purpose of this research study is to understand effects of a complementary medicine therapy, Healing Touch on quality of life and immunity of patients who are receiving treatment for breast cancer. Healing Touch is a Holistic Therapy used as an adjunct to medical treatment. The goal of Healing Touch is to restore energy and vitality to the body as a patient is receiving treatment for cancer. Treatments include light touch on specific points on the body as well as around the body, to increase well-being and support the body's ability to heal. Healing Touch has been shown to increase relaxation and well-being and to decrease anxiety, pain, and treatment side effects in a variety of illnesses including cancer. Although Healing Touch is frequently used by cancer patients along with their medical treatments, very little is understood about the effects of this treatment on the immune system. The immune system is known to be important in the body's response to fighting cancer. We are studying Healing Touch to help us understand whether or not these treatments are effective in supporting the immune system during breast cancer treatment

Aim 1. To evaluate effects of a healing touch (HT) intervention on cellular immunity among early stage breast cancer patients during radiotherapy.

Aim 2. To evaluate effects of a Healing Touch (HT) intervention on cytokines associated with radiation damage and acute skin reactions in early stage breast cancer patients during radiotherapy.

Aim 3. To evaluate the effects of a Healing Touch intervention on fatigue and mood in early stage breast cancer patients during radiation treatment.

DETAILED DESCRIPTION:
Breast cancer patients use Complementary and Alternative Medicine (CAM) in greater proportions than any other group of cancer patients. The primary reason breast cancer patients cite for use of CAM is strengthening the immune system. Healing touch (HT) is a CAM treatment frequently used by cancer patients to reduce adverse side effects of chemotherapy and radiation and to enhance immunity. HT is classified by NIH as a "biofield" therapy as its effects are proposed to be secondary to manipulation of "energy fields" around the body of a patient. A recent meta-analysis has demonstrated relatively large effects of HT on well-being and on physiological parameters, even from brief treatments. However, to date, there are no data on the effects of HT on immune function among breast cancer patients during treatment. This is particularly important as several immune parameters show long-term suppression or alteration, particularly after combined adjuvant chemotherapy and radiation among breast cancer patients. Additionally, there are no data on the effects of HT on the common side effects of breast cancer treatment which can include profound fatigue and radiation-induced skin damage. Physiological mechanisms underlying possible effects of HT are also poorly understood. This study is designed to reduce this knowledge gap by examining how HT affects cellular immune function and biomarkers related to two of the most problematic side effects of breast cancer treatment, fatigue and radiation-induced tissue damage. Effects on the subjective experience of fatigue and clinician rated skin damage will also be noted. Participants will be 42 early stage breast cancer patients who are receiving a standard course of radiotherapy following breast conservation surgery or mastectomy who have either had chemotherapy or not

The significance of the project is as follows. If positive effects are demonstrated on intermediate outcomes such as immune parameters, markers of radiation damage, and/or fatigue, follow-up studies would be warranted examining effects of HT on a) recurrence and survival, b) incidence of long term side effects of radiation, c) quality of life among breast cancer patients. Additionally, if effects of HT are demonstrated, a critical examination of putative mechanisms of action, using controls for effect of attention, expectation, and other placebo effects will be warranted.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who have received either a mastectomy or breast conservative surgery
* Diagnosis of Stage I-IIIa breast cancer,
* Receiving either chemotherapy + radiation or radiation alone

Exclusion Criteria:

* Past history of cancer
* Recurrent cancer
* Greater than Stage IIIa breast cancer
* History of immunosuppressive disorders (e.g. HIV, AIDS, hepatitis, etc.)
* On immunosuppressive medications
* On corticosteroids (e.g. Prednisone)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-07 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
NK cell activity; sTNFRII; IL-1ra; fatigue (FSI); depression (CES-D); acute skin reactions | six weeks

SECONDARY OUTCOMES:
WBC, distress (POMS), sleep quality, days of interrupted treatment | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Lutgendorf, PhD, Principal Investigator — Department of Psychology, University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Archambeau JO, Pezner R, Wasserman T. Pathophysiology of irradiated skin and breast. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1171-85. doi: 10.1016/0360-3016(94)00423-I. PMID 7713781
- [Background] Whiteside TL, Herberman RB. Role of human natural killer cells in health and disease. Clin Diagn Lab Immunol. 1994 Mar;1(2):125-33. doi: 10.1128/cdli.1.2.125-133.1994. PMID 7496932
- [Background] Jacobson JS, Verret WJ. Complementary and alternative therapy for breast cancer: the evidence so far. Cancer Pract. 2001 Nov-Dec;9(6):307-10. doi: 10.1046/j.1523-5394.2001.96001.x. No abstract available. PMID 11879333
- [Background] Menthe J. Healing touch level I notebook, 1996.
- [Background] Freel M, Hart L. Nurse's handbook of Alternative & Complementary therapies. Apringhouse, PA: Springhouse Publishing Co.: 61-82, 1999.
- [Background] Bogulawski M. Therapeutic touch: a facilitator of pain relief. Top Clin Nurs. 1980 Apr;2(1):27-37. No abstract available. PMID 6992355
- [Background] Wirth DP, Richardson JT, Eidelman WS. Wound healing and complementary therapies: a review. J Altern Complement Med. 1996 Winter;2(4):493-502. doi: 10.1089/acm.1996.2.493. PMID 9395679
- [Background] Astin JA, Harkness E, Ernst E. The efficacy of "distant healing": a systematic review of randomized trials. Ann Intern Med. 2000 Jun 6;132(11):903-10. doi: 10.7326/0003-4819-132-11-200006060-00009. PMID 10836918
- [Result] Bower JE, Ganz PA, Desmond KA, Rowland JH, Meyerowitz BE, Belin TR. Fatigue in breast cancer survivors: occurrence, correlates, and impact on quality of life. J Clin Oncol. 2000 Feb;18(4):743-53. doi: 10.1200/JCO.2000.18.4.743. PMID 10673515
- [Result] Lindley C, Vasa S, Sawyer WT, Winer EP. Quality of life and preferences for treatment following systemic adjuvant therapy for early-stage breast cancer. J Clin Oncol. 1998 Apr;16(4):1380-7. doi: 10.1200/JCO.1998.16.4.1380. PMID 9552041
- [Result] Oberst MT, Hughes SH, Chang AS, McCubbin MA. Self-care burden, stress appraisal, and mood among persons receiving radiotherapy. Cancer Nurs. 1991 Apr;14(2):71-8. PMID 2044064
- [Result] Melief CJ. Tumor eradication by adoptive transfer of cytotoxic T lymphocytes. Adv Cancer Res. 1992;58:143-75. doi: 10.1016/s0065-230x(08)60294-8. No abstract available. PMID 1532109
- [Result] Hamaoka T, Fujiwara H. Phenotypically and functionally distinct T-cell subsets in anti-tumor responses. Immunol Today. 1987;8(9):267-9. doi: 10.1016/0167-5699(87)90186-1. PMID 25344282
- [Result] Hung K, Hayashi R, Lafond-Walker A, Lowenstein C, Pardoll D, Levitsky H. The central role of CD4(+) T cells in the antitumor immune response. J Exp Med. 1998 Dec 21;188(12):2357-68. doi: 10.1084/jem.188.12.2357. PMID 9858522
- [Result] Levy SM, Herberman RB, Maluish AM, Schlien B, Lippman M. Prognostic risk assessment in primary breast cancer by behavioral and immunological parameters. Health Psychol. 1985;4(2):99-113. doi: 10.1037//0278-6133.4.2.99. PMID 4018006
- [Result] Levy S, Herberman R, Lippman M, d'Angelo T. Correlation of stress factors with sustained depression of natural killer cell activity and predicted prognosis in patients with breast cancer. J Clin Oncol. 1987 Mar;5(3):348-53. doi: 10.1200/JCO.1987.5.3.348. PMID 3546612
- [Result] Levy SM, Herberman RB, Lee J, Whiteside T, Kirkwood J, McFeeley S. Estrogen receptor concentration and social factors as predictors of natural killer cell activity in early-stage breast cancer patients. Confirmation of a model. Nat Immun Cell Growth Regul. 1990;9(5):313-24. PMID 2077396
- [Result] Tichatschek E, Zielinski CC, Muller C, Sevelda P, Kubista E, Czerwenka K, Spona J, Wolf H, Eibl MM. Long-term influence of adjuvant therapy on natural killer cell activity in breast cancer. Cancer Immunol Immunother. 1988;27(3):278-82. doi: 10.1007/BF00205452. PMID 2460239
- [Result] Morris KT, Johnson N, Homer L, Walts D. A comparison of complementary therapy use between breast cancer patients and patients with other primary tumor sites. Am J Surg. 2000 May;179(5):407-11. doi: 10.1016/s0002-9610(00)00358-5. PMID 10930491
- [Result] Wirth D. The effect of non-contact therapeutic touch on the healing rate of full thickness dermal wounds. Subtle Energies 1:1-20, 1990.
- [Result] Wirth D, Brenlan D, Levine R, Rodriguez C. The effect of complementary healing therapy on postoperative pain after surgical removal of impacted third molar teeth. Complementary Therapies in Medicine 2:187-192, 1994.
- [Result] Wirth D, Richardson J, Eidelman W, O'Malley A. Full thickness dermal wounds treated with non-contact therapeutic touch: A replication and extension. Complemenatary Therapies in Medicine 1:127-132, 1993.
- [Result] Wirth D, Barret M, Eidelman W. Non-contact therapeutic touch and wound re-epithelialization: An extension of previous research. Complementary Therapies in Medicine 2:187-192, 1994.
- [Result] Quinn JF. Therapeutic touch as energy exchange: testing the theory. ANS Adv Nurs Sci. 1984 Jan;6(2):42-9. doi: 10.1097/00012272-198401000-00007. PMID 6322674
- [Result] Keller E, Bzdek VM. Effects of therapeutic touch on tension headache pain. Nurs Res. 1986 Mar-Apr;35(2):101-6. PMID 3633503